CLINICAL TRIAL: NCT06304064
Title: Open-Label Extension of the Halt Cardiomyopathy Progression in Duchenne (HOPE-Duchenne) Trial (CAP-1002-DMD-03)
Brief Title: Halt cardiomyOPathy progrEssion in Duchenne (HOPE-OLE)
Acronym: HOPE-OLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capricor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAP-1002-DMD-03
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Cardiomyopathy; Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Allogeneic Cardiosphere-Derived Cells (CAP-1002) (Experimental): All participants who were randomized to the Usual Care Treatment Group and completed 12 months of follow-up in the HOPE-Duchenne trial (NCT02485938), will receive CAP-1002 intravenous infusion on Day 1 and at Month 3 in the current study.
  Interventions: Biological: Allogeneic Cardiosphere-Derived Cells (CAP-1002)

INTERVENTIONS:
Biological: Allogeneic Cardiosphere-Derived Cells (CAP-1002) — Intravenous infusion delivery of Allogeneic Cardiosphere-Derived Cells (CAP-1002; 75 million CDCs)
  Other Names: CAP-1002

SUMMARY:
This Phase 2, multi-center, open-label extension trial will provide CAP-1002 to participants who were randomized to the Usual Care treatment group of the HOPE-Duchenne study (NCT02485938) and completed 12 months of follow-up.

The trial will assess the safety and efficacy of two intravenous administrations of CAP-1002, each separated by three months.

DETAILED DESCRIPTION:
Participants with documented enrollment in the Usual Care treatment group of the HOPE-Duchenne study and completion of study follow-up through Month 12 were eligible for this study.

Participants will undergo a targeted screening during a 30-day screening period, eligible subjects will then undergo baseline safety and efficacy assessments on Day 1 prior to their first infusion of CAP-1002.

All CAP-1002 infusions will be conducted in an outpatient setting at the investigative site on Day 1 and at Month 3. Participants will be observed in the outpatient setting for at least two hours post-infusion and then discharged the same day if medically cleared by the site Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Documented enrollment in the Usual Care Treatment Group of the HOPE-Duchenne trial and completion of trial follow-up through Month 12.
2. Willing and able to provide informed consent to participate in the trial if greater than or equal to (>=) 18 years of age, and assent with parental or guardian informed consent if less than (<) 18 years of age.
3. Adequate venous access for intravenous CAP-1002 infusions and routine blood collections in the judgement of the Investigator.
4. Assessed by the Investigator as willing and able to comply with the requirements of the trial.

Exclusion Criteria:

1. Left ventricular ejection fraction (LVEF) < 35 percent (%) within 6 months of screening.
2. Planned or likely major surgery in the next 6 months after planned first infusion.
3. Risk of near-term respiratory decompensation in the judgment of the investigator, or the need for initiation of non-invasive ventilator support as defined by serum bicarbonate >= 29 millimoles per liter (mmol/L) at screening.
4. History of non DMD-related chronic respiratory disease including, but not limited to, asthma, bronchitis, and tuberculosis.
5. Acute respiratory illness within 30 days prior to screening.
6. Known hypersensitivity to dimethyl sulfoxide (DMSO) or bovine products.
7. Treatment with investigational product <= 6 months prior to first infusion.
8. History, or current use, of drugs or alcohol that could impair ability to comply with participation in the trial.
9. Inability to comply with the investigational plan and follow-up visit schedule for any reason, in the judgment of the investigator.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Awadalla, Study Director — Capricor Inc.
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Cincinnati Children's Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Allogeneic Cardiosphere-Derived Cells (CAP-1002): All participants who were randomized to the Usual Care Treatment Group and completed 12 months of follow-up in the HOPE-Duchenne trial (NCT02485938) and received CAP-1002 intravenous infusion on Day 1 and at Month 3 in the current study.
Period: Overall Study
Arm/Group | Allogeneic Cardiosphere-Derived Cells (CAP-1002)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- CAP-1002: All participants who were randomized to the Usual Care Treatment Group and completed 12 months of follow-up in the HOPE-Duchenne trial (NCT02485938), and received CAP-1002 intravenous infusion on Day 1 and at Month 3 in the current study.
Arm/Group | CAP-1002
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.8 (2.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Acute Respiratory Decompensation
Description: Acute respiratory decompensation is defined as an unexplained rapid deterioration of the participant's condition with increasing shortness of breath requiring oxygen supplementation. Acute respiratory decompensation within 2 hours following investigational product (IP) administration will be reported.
Time Frame: 2 hours post-dose on Day 1 and Month 3
Population: Analysis was performed on safety population that included all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | CAP-1002
Number analyzed (Participants) | 8
Participants
  Day 1 | 0
  Month 3 | 0

2. Primary Outcome: Number of Participants With Hypersensitivity Reactions
Description: Hypersensitivity reaction is defined as a clinical syndrome including, but not limited to, fever, leukocytosis, or rash with onset <= 2 hours post-infusion and lasting < 24 hours, in the absence of clinical signs of concomitant infection.
Time Frame: From Day 1 up to Month 6
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAP-1002
Number analyzed (Participants) | 8
Participants | 1

3. Primary Outcome: All-cause Mortality
Description: Number of deaths due to any cause will be reported.
Time Frame: From Day 1 up to Month 6
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAP-1002
Number analyzed (Participants) | 8
Participants | 0

4. Primary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) Related to Investigational Product or Administration and Serious Adverse Events (SAEs)
Description: An adverse events (AEs) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. TEAEs are defined as AEs occurring after the initiation of the IV catheter placement for the initial dose of IP. TEAEs related to investigational product or administration are reported for this outcome measure. A SAE is defined as an AE that results in any of the following outcomes: Death; life-threatening adverse event; Inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; congenital anomaly/birth defect.
Time Frame: From Day 1 up to Month 6
Population: Analysis was performed on safety population.
Measure: Number; unit: number of events
Arm/Group | CAP-1002
Number analyzed (Participants) | 8
number of events
  TEAEs | 11
  TESAEs | 1

5. Primary Outcome: Number of Participants With Immune Sensitization Syndrome
Description: Immune sensitization syndrome shall be defined as: (a) clinical signs and symptoms consistent with systemic inflammation (e.g., fever, leukocytosis, rash, or arthralgia) with onset >= 24 hours post infusion and the absence of clinical signs of concomitant infection, and (b) elevation of anti-human leukocyte antigen (HLA) antibodies against the donor cells (i.e., DSAs), detected <= 30 days following onset of syndrome, of (i) >= 2000 mean fluorescent intensity (MFI) if baseline MFI <= 1000, or (ii) >= 2 times baseline otherwise.
Time Frame: From Day 1 up to Month 6
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAP-1002
Number analyzed (Participants) | 8
Participants | 0

ADVERSE EVENTS:
Time Frame: From Day 1 up to Month 6
Arm/Group | CAP-1002
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAP-1002 (N=8)
Anaphylactic Reaction (Immune system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAP-1002 (N=8)
Nasopharyngitis (Infections and infestations) | 3
Oesophageal Ulcer (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 2
Drug Eruption (Skin and subcutaneous tissue disorders) | 1
Tachycardia (Cardiac disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Eye Pain (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Onychomycosis (Infections and infestations) | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT06304064/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT06304064/SAP_001.pdf